CLINICAL TRIAL: NCT06316310
Title: The Effect and Safety of Acupoint Thread Embedding on Over-weight and Obesity Treatment : A Randomized, Single-Blind, Sham- Controlled Study
Brief Title: Effect of Acupoint Thread Embedding on Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XSF20240312
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-03

CONDITIONS: Obesity
Keywords: Acupoint Thread Embedding; Sham Acupoint Thread Embedding; Obesity; Randomized Controlled Trial
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: All eligible participants will be randomly assigned into two group at a ratio of 1:1, the Acupoint Thread Embedding group and the Sham Acupoint Thread Embedding group (the control group).
  group).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupoint Thread Embedding group+health education (Active Comparator): Acupuncture thread embedding (ATE), extension and development of acupuncture therapy, which emerged in mid 1950s, is an acupoint stimulation technique which sterile biodegradable threads (such as polydioxanone (PDO) threads) are inserted into acupuncture points, by using hollow core embedding needles. The aim of this therapy is provide long term stimulation of acupoints, making this technique one of the most commonly used methods for treating obesity.
  Interventions: Other: acupoint thread embedding
- Sham Acupoint Thread Embedding group+health education (Sham Comparator): Sham acupoint thread embedding method in this study is set as the Sham acupoint thread embedding manipulated at the same main acupoints won't be put into trocar and de qi sensation will not be obtained.
  The aim of the sham acupoint thread embedding is to eliminate the possible placebo effect of ATE treatment.
  Interventions: Other: acupoint thread embedding

INTERVENTIONS:
Other: acupoint thread embedding — Acupoint embedding therapy:Main acupoints: Shangguan (CV-13), Xiaguan (CV-10), Tianshu (ST-25), Daheng (SP-15), Fenglong (ST-40), Qihai (CV-6), Zhongguan (CV-12), Zusanli (ST-36), Quchi (LI-11), Guanyuan (CV-4), Wailing (ST-26), Daju (ST-27), Shuidao (ST-28), Daimai (GB-26), Liangmen (ST-21), Ashi acupoints , where local fat accumulation in the abdomen. Methods of operation: With the patient in the prone position and all acupoints routinely sterilized, the acupuncturist will use sterile forceps to insert a 3-0 × 2-cm poly-p-dimethyl-hydroxy-oxazolone (PDO) thread into the tip of the #6 (0.6 mm × 60 mm) disposable embedded thread needle. The tissue around the area of the acupuncture point will be lifted with the thumb and forefinger of the non-dominant hand and the needle will be inserted into the acupuncture point to a depth of 1.5 cm with the dominant hand. Each treatment will last maximum of 10 minutes and the intervention will be repeated every 2 weeks for a total of 6 sessions.
  Other Names: sham acupoint thread embedding

SUMMARY:
The investigators describe a protocol for a randomized controlled trial to find out the effect and safety of acupoint thread embedding on losing weight in obese patients.

DETAILED DESCRIPTION:
Obesity refers to a complex chronic disease in which there is excessive accumulation of body fat. As of 2016, there were more than 650 million obese people worldwide, and it is expected to reach 1.12 billion by 2030, with at least 2.8 million deaths due to obesity each year, according to surveys. In Europe, 60 percent of the population is already overweight or obese. The incidence of obesity is also increasing rapidly in China, with a recent report by The Lancet showing that the number of obese people in China has reached 85 million, making it the country with the highest number of obese people in the world. In 2002, the China Obesity Task Force recommended threshold value to define overweight as Body Mass Index (BMI) of ≥ 24 kg/m2, a waist circumference (WC) ≥of 85 cm for men and a WC ≥ 80 cm for women, or a Waist-to-Hip Ratio (WHR) of ≥ 0.9 for men and a WHR ≥ 0.8 for women, and to define obesity as a BMI ≥ 28 kg/m2. Studies have shown that Asian populations have higher health risks at the same BMI and WC levels due to the distribution of adipose tissue. Acupoint thread embedding is a widely recognized therapy to lose weight in clinical practice.But there are some doubts about the effectiveness of acupoint thread embedding versus sham acupoint thread embedding in treating obesity due to its lack of medical evidence.

This randomized placebo-controlled clinical trial is aimed to investigate the effect and safety of acupoint thread embedding (ATE) in obese patients. The investigators designed a protocol for a randomized controlled trial, in which 132 eligible patients will be randomly assigned to one of the two groups: the ATE group (receiving ATE treatment with health education) and the sham acupoint thread embedding (SATE) group (receiving SATE treatment with health education). A total of 6 sessions of interventions will be given for consecutive 12 weeks, followed by 12 weeks follow-up period. Each session of ATE or SATE treatment will last for about 30 minutes. The primary outcome is the change of the body mass index (BMI) at week 12. The secondary outcomes include the change of patient's body weight and body circumference, results from the blood tests (FBG, LDL-C, HDL-C, TG and TC), the abdominal visceral fat tissue thickness scanned by FibroScan, data collected from the body composition analyzer, and the scores of the impact of weight on quality of life (IWQOL-Lite), the well-being index (WHO-5), visual analog scale (VAS) of appetite and hamilton anxiety scale(HAMA). All adverse effects will be accessed by the treatment emergent symptom scale (TESS) from baseline to the follow-up period. The body weight and circumferences，BMI，IWQOL-Lite, WHO-5, VAS, and the HAMA, will be calculated at baseline, week 6, week 12, and week 24. blood tests，FibroScan and the body composition analyzer's data will be calculated at baseline，week 12 and week24. All patients will be provided with the same health education brochure to choose more beneficial personalized lifestyle during the 12-week intervention period.

All analyses will be performed on the intention-to-treat (ITT) population of participants who have at least one treatment. Missing data will be handled using the multiple imputation method, on the assumption that values at each time point follow a specific distribution calculated by the computer software R V.3.5. The primary outcome is the change of the body mass index (BMI) at week 12. Linear mixed effects models will be used for analyses with the use of the statistical software SPSS V.29.0. The t-test will be used to compare the measurement data between either two groups from the baseline to follow-up; the rank sum test will be used for ranked data while the Chi-squared test will be used to analyze categorical data. The significance level that will be used for statistical analysis with 2-tailed testing will be 2.5%. Data values will mainly be presented as Mean±SD. The findings from this trial will help further explore the efficacy and safety of ATE on losing weight for patients with obesity, as well as determine the differences between the ATE and SATE treatment.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18~45 years old;
* BMI≥24.0 kg/m2；
* WC≥80cm ; recommended BMI and WC threshold value to define overweight in China;
* Stable weight change (increase or decrease of ≤4 kg) within 3 months prior to the start of the test;
* Agree to participate in the trial and sign a written informed consent form;

Exclusion Criteria:

* Secondary obesity caused by drugs, or neuro-endocrine-metabolic disorders (such as thalamic disease, hypopituitarism, etc.);
* History of bariatric surgery (gastric reduction, liposuction, etc.);
* Are taking medications that may affect the results of the trial (weight):
* Severe ulcers, abscesses, skin infections, etc. at the acupuncture site;
* Severe heart, brain, lung, liver and kidney insufficiency, hematopoietic system disease or other serious diseases;
* Participated in other clinical medical trial studies in the past 1 month;
* History of acupoint thread embedding in the past 6 months;
* Alcoholism, drug abuse, or smoking (change in smoking habits within the past 2 months or a plan to quit smoking during the study period);
* Pregnant and lactating women.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | week12
  one of the criteria for evaluating the body weight and health status of a person. BMI = weight (kg)/height (m)2. Each subject will be provided with a free Bluetooth Internet-enabled scale to monitor their weight at regular intervals, and the researcher will be able to access the data from the backend.

SECONDARY OUTCOMES:
Change in body weight | week0, week6, week12, week24
  The change in body weight at the end of the intervention compared to the baseline.
Body Mass Index (BMI) | week0, week6, week24
  one of the criteria for evaluating the body weight and health status of a person. BMI = weight (kg)/height (m)2. Each subject will be provided with a free Bluetooth Internet-enabled scale to monitor their weight at regular intervals, and the researcher will be able to access the data from the backend
Changes in body circumference | week0, week6, week12, week24
  Waist circumference (WC), hip circumference (HC), waist-hip ratio (WHR), waist-height ratio (WHtR), and the average value of the changes in each circumference at the end of the intervention were calculated compared with the baseline. WHR=WC/HC; WHtR=WC/height .
Body composition analysis | week0, week12, week24
  Evaluating changes in body fat percentage or composition by using bioelectrical impedance analysis (BIA) device (InBody770; Biospace, Seoul, Korea)., which allows for high-density body composition measurements, including muscle mass, body water content, body fat percentage, visceral fat grade, and other body components, by bioelectrical impedance analysis.
Changes in liver fat content | week0, week12, week24
  Liver fat changes are quantitatively calculated with FibroScan.
Fasting blood glucose (FPG) | week0, week12, week24
  glucose concentration in the blood in the early morning fasting, which can reflect the function of pancreatic β-cells,HOMA-IR, Insulin level.
Blood lipid profile | week0, week12, week24
  including Low-density Lipoprotein (LDL), High density lipoprotein (HDL), triglyceride (TG), cholesterol (TC), reflects the lipid metabolism within the body.
Impact of Weight on Quality-of-Life Scale (IWQOL-Lite) | week0, week6, week12, week24
  a 31-item self-report scale consisting of a total score and individual scores on 5 dimensions, i.e., physical functioning, self-esteem, sexuality, public stress, and work, to assess the quality of life of obese patients
Well-Being Index (WHO-5) | week0, week6, week12, week24
  shot, self-administered subjective measure of well-being over the last two weeks. It consists of 5 positively worded item that is rated on 0-6 which is 0 means at no time and 5 is all the time.
Visual analog scale (VAS) of appetite | week0, week6, week12, week24
  This method relies on a line segment of 100 mm or 150mm in length, with the two ends pointing to "I have no appetite at all" and "I have a very good appetite" respectively. Subjects mark the line according to their level of appetite. The patient was determined to have a reduced appetite if the measured line segment was <50 mm or 70 mm.
Hamilton Anxiety Scale (HAMA) | week0, week6, week12, week24
  The CCMD-3 Chinese Diagnostic Criteria for Mental Disorders lists it as an important diagnostic tool for anxiety disorders, and is often used clinically as the basis for the diagnosis and degree classification of anxiety disorders. The total score can better reflect the severity of anxiety symptoms, and can be used to evaluate the severity of anxiety symptoms in patients with anxiety and depressive disorders and evaluate the effects of various drugs and psychological interventions. According to the information provided by the Chinese scale collaboration group: the total score is ≥ 29 points, which may be severe anxiety; ≥ 21 points, there must be significant anxiety; ≥ 14 points, there is definitely anxiety; More than 7 points, there may be anxiety; If the score is less than 7, there are no anxiety symptoms.
Adverse effects | week6, week12, week24
  Any adverse event (described as unfavourable or unintended signs, symptoms or diseases occurring during the trial) related to the intervention will be reported by patients and practitioners and accessed by the Treatment Emergent Symptom Scale (TESS) which is used as an associated indicator to mainly evaluate the safety of acupoint thread embedding treatment in this trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data in this trial will be publicly available from the corresponding author upon reasonable request. All data and the protocol will be available after publication in peer-reviewed international journals for 3 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All data and the protocol will be available after publication in peer-reviewed international journals for 3 years.
Access Criteria: The data in this trial will be publicly available from the corresponding author upon reasonable request.